CLINICAL TRIAL: NCT04016220
Title: Nebulized Budesonide Combined With Systemic Corticosteroid in Acute Severe Asthma Managed in the Emergency Department: A Randomized Controlled Trial
Brief Title: Nebulized Budesonide Combined With Systemic Corticosteroid in Acute Severe Asthma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Soudani MARGHLI, MD, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Monastir
Record Dates: First submitted 2019-05-29; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Acute Asthma
Keywords: asthma; budesonide; nebulized; adult
MeSH Terms: conditions — Asthma | interventions — Budesonide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: senior ED and patient do not know the randomization group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Budesonide group (Experimental): The experimental group received a first nebulization of 5 mg of terbutaline(solution of 5mg/ 2 ml ) in association with 0.5 mg of ipratropium bromide (solution of 0.5 mg/ 2 ml) and 0.5 mg of budesonide (solution of 0.5 mg/2 ml) followed by repetitive nebulization of 5 mg of terbutaline with 0.5 mg of budesonide at 20, 40, 60 and 120 min. All patients received hydrocortisone hemisuccinate (100 mg i.v.) and O2 (7 l/ min) via a nebulizer.
  Interventions: Drug: Budesonide
- normal saline (Placebo Comparator): The control group received a nebulization of 2 ml normal saline at baseline, 20, 40, 60 and 120 min as placebo comparator in association with nebulized terbutaline . All patients received hydrocortisone hemisuccinate (100 mg i.v.) and O2 (7 l/ min) via a nebulizer.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Budesonide — first nebulization of 0.5 mg of budesonide in association with terbutaline and ippratropium bromide followed by repetitive nebulization of 5 mg of terbutaline with 0.5 mg of budesonide at 20, 40, 60 and 120 min.
  Arms: Budesonide group
Drug: normal saline — first nebulization of 2ml of normal saline as placebo comparator in association with terbutaline and ippratropium bromide followed by repetitive nebulization of 5 mg of terbutaline with 2 ml of normal saline at 20, 40, 60 and 120 min.
  Arms: normal saline

SUMMARY:
Our study is a prospective double-blind randomized study performed in the Emergency Department (ED). The objective of our study was to demonstrate the additive effect of high and repeated doses of inhaled budesonide combined with the standard treatment of acute asthma in adult managed in the ED

DETAILED DESCRIPTION:
Patients were included in a double-blind, randomized into one of two groups. The experimental group received a first nebulization of 5 mg of terbutaline (Bricanyl®, AstraZeneca : solution of 5mg/ 2 ml ) in association with 0.5 mg of ipratropium bromide (Ipratropium®, AGUETTANT, solution of 0.5 mg/ 2 ml) and 0.5 mg of budesonide (Pulmicort®, AstraZeneca, solution of 0.5 mg/2 ml) followed by repetitive nebulization of 5 mg of terbutaline with 0.5 mg of budesonide at 20, 40, 60 and 120 min. The control group received a first nebulization of 5 mg of terbutaline in association with 0.5 mg of ipratropium bromide and 2 ml of normal saline followed by a repetitive nebulization of 5 mg de terbutaline with 2 ml of normal saline at 20, 40, 60 and 120 min (Figure 1). The placebo and the budesonide were prepared by the pharmacist. All patients received hydrocortisone hemisuccinate (100 mg i.v.) and O2 (7 l/ min) via a nebulizer (Mini nebulizer 40-115510; Peters, France).

Measure The following parameters were measured in each patient immediately before starting the treatment and at 30 minute intervals for 3 hours after presentation: peak expiratory flow (PEF), respiratory rate (RR), heart rate (HR), dyspnea scale, systolic and diastolic blood pressure. PEF was measured with peak flow meter (mini-Wright; Clement Clarke; Harlow, UK). The highest of three values was recorded. HR was measured from continuous monitor. Dyspnea was assessed by the patient's own sensation of respiratory difficulty with a value assigned on a scale of 0 to 3, in which 0 denoted absent, 1 mild, 2 moderate, and 3 severe. At the end of the treatment, the patient was asked to indicate the presence or absence of each of five symptoms: palpitations, tremor, anxiety, headache, and dry mouth. Also, an interviewer determined the duration of symptoms before presentation, which specifically included how long the patient had been wheezing and shorter of breath than usual; a decline in the PEF, if available, was considered. The occurrence of a worsening of ventilator status requiring mechanical ventilation led to interrupt the study protocol. The decision to discharge or admit a patient was made at the end of the protocol (180 minutes) by a senior ED staff without knowledge of previous patient group allocation. Although some patients met discharge criteria during the study, none were discharged until the end of the protocol. Patients were discharged from the ED according to the following criteria: if accessory-muscle use disappeared, if wheezing was judged minimal to completely resolved, if they were free of dyspnea, and if PEF was more than 60% of predicted value. Physicians prescribed oral prednisone (40 mg for 7 days) for all discharged patients.

ELIGIBILITY:
Inclusion Criteria:

* acute asthma
* peak expiratory flow (PEF) rate less than 50% of predicted value
* one or more of the following features were present: accessory muscle activity, a heart rate greater than 110 beats/minute, a respiratory rate greater than 25 breaths/minute, a limited ability to speak
* written informed consent obtained

Exclusion Criteria:

* temperature higher than 38°C
* history of cardiac, hepatic, renal, or other medical disease
* pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
admission rate | 3 hours
  The decision to discharge or admit a patient was made at the end of the protocol (180 minutes)

SECONDARY OUTCOMES:
Peak expiratory flow | 3 hours
  Peak expiratory flow (L/min) was measured in each patient immediately before starting the treatment and at 30 minute intervals for 3 hours after presentation.
respiratory rate was measured in each patient immediately before starting the treatment and at 30 minute intervals for 3 hours after presentation. | 3 hours
  respiratory rate
dyspnea scale | 3 hours
  Dyspnea was assessed by the patient's own sensation of respiratory difficulty with a value assigned on a scale of 0 to 3, in which 0 denoted absent, 1 mild, 2 moderate, and 3 severe. was measured in each patient immediately before starting the treatment and at 30 minute intervals for 3 hours after presentation:
Hear rate | 3 hours
  Heart rate was measured in each patient immediately before starting the treatment and at 30 minute intervals for 3 hours after presentation.
tremor | 3 hours
  incidence of tremor
dry mouth | 3 hours
  incidence of dry mouth
palpitation | 3 hours
  incidence of palpitation
headache | 3 hours
  incidence of headache

CONTACTS AND LOCATIONS:
Overall Officials: Soudani Marghli, Professor, Principal Investigator — University of Monastir Tunisia
Locations (1):
- University of Monastir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guttman A, Afilalo M, Colacone A, Kreisman H, Dankoff J. The effects of combined intravenous and inhaled steroids (beclomethasone dipropionate) for the emergency treatment of acute asthma. The Asthma ED Study Group. Acad Emerg Med. 1997 Feb;4(2):100-6. doi: 10.1111/j.1553-2712.1997.tb03714.x. PMID 9043535
- [Background] Bateman ED, Fairall L, Lombardi DM, English R. Budesonide/formoterol and formoterol provide similar rapid relief in patients with acute asthma showing refractoriness to salbutamol. Respir Res. 2006 Jan 24;7(1):13. doi: 10.1186/1465-9921-7-13. PMID 16433920
- [Result] Rodrigo GJ. Comparison of inhaled fluticasone with intravenous hydrocortisone in the treatment of adult acute asthma. Am J Respir Crit Care Med. 2005 Jun 1;171(11):1231-6. doi: 10.1164/rccm.200410-1415OC. Epub 2005 Mar 11. PMID 15764724
- [Derived] Marghli S, Bouhamed C, Sghaier A, Chebbi N, Dlala I, Bettout S, Belkacem A, Kbaier S, Jerbi N, Bellou A. Nebulized budesonide combined with systemic corticosteroid vs systemic corticosteroid alone in acute severe asthma managed in the emergency department: a randomized controlled trial. BMC Emerg Med. 2022 Jul 23;22(1):134. doi: 10.1186/s12873-022-00691-9. PMID 35870902